CLINICAL TRIAL: NCT05389449
Title: A Long-term Extension (LTE) Study to Characterize the Safety and Efficacy of Danicopan as an Add-on Therapy to a Complement Component 5 Inhibitor (C5i) in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Previously Treated With Danicopan in an Alexion-sponsored Clinical Study
Brief Title: A Long-term Safety and Efficacy Study of Danicopan as an Add-on Therapy to Complement Component 5 Inhibitor (C5i) in Participants With PNH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN2040-PNH-303
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Paroxysmal Nocturnal Hemoglobinuria (PNH); Extravascular Hemolysis (EVH); Factor D inhibitor; Complement; Danicopan; ALXN2040; C5 inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis | interventions — danicopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Danicopan (Experimental): Participants will receive their last dose of danicopan from the parent study the night prior to Day 1 of this LTE study and will continue daily treatment with danicopan together with their background C5i therapy.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Oral tablet
  Other Names: ALXN2040, ACH-0144471

SUMMARY:
This is a single-arm long-term extension study that will enroll participants with PNH who have completed participation in Alexion-sponsored clinical studies with danicopan as an add on therapy to a C5i.

DETAILED DESCRIPTION:
The total duration of the study will be up to 3 years. Eligible participants must complete all study assessments on the parent protocol before starting this study. All participants entering this study will receive danicopan as an add-on to a background C5i therapy. The only allowed C5i therapies are eculizumab and ravulizumab.

ELIGIBILITY:
Key Inclusion Criteria:

* All participants who completed their participation in an Alexion sponsored clinical study with danicopan as an add on to a C5i treatment.
* Patient is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
* Documentation of vaccination for Neisseria meningitidis: All participants must be revaccinated as per national vaccination guidelines or local practice for vaccination use with complement inhibitors.

Key Exclusion Criteria:

* Any medical condition (for example, cardiac, pulmonary, renal, oncologic, or psychiatric) that, in the opinion of the Investigator, might interfere with participation in the study, pose any added risk to the participant, or confound the assessment of the participant.
* Patient has been permanently discontinued from danicopan in the parent study for any reason other than enrollment into this LTE study.
* Female participants who are pregnant, breastfeeding, or intending to conceive during the course of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Participants Experiencing Treatment-emergent Adverse Events (TEAEs) And Serious TEAEs | Up to 3 years

SECONDARY OUTCOMES:
Change In Hemoglobin Values | Up to 3 years
Proportion of patients with Hgb increase ≥ 2g/dL in the absence of transfusion over time | Up to 3 years
Change In Absolute Reticulocyte Count | Up to 3 years
Change In Lactate Dehydrogenase (LDH) | Up to 3 years
Proportion Of Participants With LDH ≤ 1.5 × Upper Limit Of Normal | Up to 3 years
Proportion Of Participants With Transfusion Avoidance | Up to 3 years
Change In Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scores | Up to 3 years
  Total scores range from 0 to 52, with higher scores indicating better QoL.
Change In The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 Scale (QLQ-C30) Scores | Up to 3 years
  Thirty questions related to QoL, with the first 28 questions scored on a 4-point scale (1 = not at all to 4 = very much) and the final 2 questions that probe the participant's overall health and QoL scored on a scale of 1 (very poor) to 7 (excellent).
Participants Experiencing TEAEs Leading To Discontinuation | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (44):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Kansas City, Missouri
  - Research Site, Long Island City, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Dallas, Texas
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
- Research Site, Toronto, Ontario, Canada
- Research Site, Brno, Czechia
- France (4):
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Israel (2):
  - Research Site, Haifa
  - Research Site, Jerusalem
- Italy (6):
  - Research Site, Avellino
  - Research Site, Bassano del Grappa
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Reggio Calabria
  - Research Site, Roma
- Japan (5):
  - Research Site, Bunkyō City
  - Research Site, Kyoto
  - Research Site, Osaka
  - Research Site, Shibuya-ku
  - Research Site, Tsukuba
- Malaysia (3):
  - Research Site, Kota Kinabalu
  - Research Site, Kuching
  - Research Site, Miri
- Research Site, Gdansk, Poland
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (4):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Majadahonda
  - Research Site, Seville
- Research Site, Bangkok, Thailand
- United Kingdom (3):
  - Research Site, Airdrie
  - Research Site, Leeds
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR